CLINICAL TRIAL: NCT07312825
Title: Postoperative Analgesic Efficacy of Combined Fascial Plane Blocks After Gynecologic Oncologic Surgery
Brief Title: Effectiveness of Combined Fascial Plane Blocks for Postoperative Pain in Gynecologic Oncology Surgery
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayşe Menekşe Çakır, Doctor of Anesthesiology, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: FASIALBLOCKJinekoOnkoAnj
Record Dates: First submitted 2025-04-07; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-04

CONDITIONS: Gynecologic Cancers; Postoperative Pain Management
Keywords: Fascial Plane Blocks for postoperative Analgesia (TAP Block, QLB, RSB); Gynecologic Oncology Surgery; Postoperative Analgesia
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: TAP Block Only Group: Patients who received only Transversus Abdominis Plane (TAP) block as part of routine anesthesia practice. No additional regional block was performed.
  Interventions: Other: Group 1:The Transversus Abdominis Plane (TAP) block
- Group 2: TAP + QLB Combination: Patients who received both TAP block and Quadratus Lumborum Block (QLB) as part of standard clinical anesthesia management.
  Interventions: Other: Group 2: TAP Block + Quadratus Lumborum Block (QLB)
- Group 3: TAP + RSB Combination: Patients who received both TAP block and Rectus Sheath Block (RSB) as part of standard clinical anesthesia management.
  Interventions: Other: Group 3: TAP Block + Rectus Sheath Block (RSB)

INTERVENTIONS:
Other: Group 1:The Transversus Abdominis Plane (TAP) block — Patients who received only Transversus Abdominis Plane (TAP) block as part of routine clinical anesthesia practice. No study-assigned intervention or randomization was performed. Data were collected prospectively from standard anesthesia records.
  Groups: Group 1: TAP Block Only Group
Other: Group 2: TAP Block + Quadratus Lumborum Block (QLB) — Patients who received TAP block combined with Quadratus Lumborum Block (QLB) during routine anesthesia management. This block combination was chosen by the attending anesthesiologist as part of standard care, not assigned by the study.
  Groups: Group 2: TAP + QLB Combination
Other: Group 3: TAP Block + Rectus Sheath Block (RSB) — Patients who received TAP block combined with Rectus Sheath Block (RSB) as part of routine anesthesia practice. The block technique was performed according to clinical judgment, not as part of a study intervention.
  Groups: Group 3: TAP + RSB Combination

SUMMARY:
The goal of this prospective observational study is to compare the effectiveness of different postoperative analgesic techniques in patients undergoing major abdominal surgery for gynecologic oncology.

The main question is whether the combination of TAP block with Quadratus Lumborum Block (QLB) or Rectus Sheath Block (RSB) provides superior pain relief compared to TAP block alone.

All blocks were performed as part of routine clinical anesthesia practice according to the attending anesthesiologist's judgment. No randomization, allocation, or study-directed intervention was performed.

Patients were classified into three groups based on the block type they received during standard care:

Group 1: TAP Block Only

Group 2: TAP + QLB Combination

Group 3: TAP + RSB Combination

Postoperative data, including pain scores (VAS), opioid consumption, sedation level, heart rate, blood pressure, nausea/vomiting, and length of hospital stay, were collected prospectively.

The study aims to determine which block combination provides the best postoperative pain control and recovery profile in patients undergoing gynecologic oncology surgery.

DETAILED DESCRIPTION:
This study is a prospective observational research designed to evaluate the postoperative analgesic effectiveness of different combinations of fascial plane blocks in patients undergoing gynecologic oncology surgery.

All blocks (Transversus Abdominis Plane [TAP] block, Quadratus Lumborum Block [QLB], and Rectus Sheath Block [RSB]) were performed as part of routine clinical anesthesia practice according to the attending anesthesiologist's preference.

No intervention, randomization, or protocol-directed procedure was applied for research purposes. After data collection, patients were classified into three groups based on the block type they had received in standard care:

TAP block only

TAP + QLB combination

TAP + RSB combination

The study prospectively compared postoperative pain scores (VAS), opioid consumption, time to mobilization, bowel function recovery, and length of hospital stay among these groups to determine the most effective analgesic strategy within routine practice.

This observational design reflects real-world anesthesia management and does not involve any experimental or interventional component.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older.
* ASA physical status I-IV.
* Scheduled for major gynecologic oncology surgery (endometrial cancer, ovarian tumor, or cytoreductive surgery).
* Undergoing general anesthesia.
* Planned postoperative abdominal fascial plane block for pain management (TAP, TAP + QLB, or TAP + RSB).
* Able to provide written informed consent.

Exclusion Criteria

* Refusal to participate or inability to provide informed consent.
* Emergency surgery.
* Known allergy or contraindication to local anesthetics.
* Infection at the block site.
* Coagulopathy or anticoagulant use that contraindicates regional anesthesia.
* Pre-existing chronic pain conditions or chronic opioid use.
* Severe hepatic or renal insufficiency.
* Cognitive impairment that prevents reliable pain assessment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult female patients who are undergoing elective major abdominal surgery due to gynecologic cancer (e.g., endometrial cancer, ovarian cancer, debulking surgery). Participants will be aged 18 years and older, and only those with ASA I-IV status who are deemed fit for surgery will be included.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Total Morphine Consumption | Within 24 hours after surgery
  Total amount of morphine (mg) administered to the patient within the first 24 hours after surgery for postoperative analgesia. Morphine use will be recorded from patient-controlled analgesia (PCA) device data or medical records.

SECONDARY OUTCOMES:
Postoperative pain intensity (VAS score) | 0-24 hours postoperatively; VAS score (0-10)
  Pain intensity will be evaluated using the Visual Analog Scale (VAS; 0 = no pain, 10 = worst pain) at 0 min, 15 min, 2 hr, 6 hr, 12 hr, and 24 hr postoperatively.
Incidence of postoperative nausea and vomiting | Time Frame: 0-24 hours postoperatively
  Number of patients experiencing postoperative nausea and/or vomiting within the first 24 hours.
Time to first gas or stool passage | From the end of surgery up to postoperative 72 hours
  Time from the end of surgery to the first postoperative bowel movement or passage of gas.
Time to mobilization | From the end of surgery up to postoperative 72 hours
  Time from the end of surgery to the first postoperative ambulation.
Time to oral intake | From the end of surgery up to postoperative 72 hours
  Time from the end of surgery to the first postoperative oral feeding
Length of hospital stay | From surgery to hospital discharge (up to 10 days) Unit of Measure:Days
  Total duration of hospitalization after surgery.
Intensive care unit (ICU) length of stay | From surgery to hospital discharge (up to 3 days) Unit of Measure: Days
  Total duration of postoperative stay in the intensive care unit.

OTHER OUTCOMES:
1.Sedation Level (Ramsey Sedation Score) | 0-24 hours after surgery
  Sedation level evaluated using the Ramsey Sedation Scale at multiple postoperative time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Yu S, Wen Y, Lin J, Yang J, He Y, Zuo Y. Combined rectus sheath block with transverse abdominis plane block by one puncture for analgesia after laparoscopic upper abdominal surgery: a randomized controlled prospective study. BMC Anesthesiol. 2024 Feb 9;24(1):58. doi: 10.1186/s12871-024-02444-6. PMID 38336613
- [Result] Zhu JL, Wang XT, Gong J, Sun HB, Zhao XQ, Gao W. The combination of transversus abdominis plane block and rectus sheath block reduced postoperative pain after splenectomy: a randomized trial. BMC Anesthesiol. 2020 Jan 23;20(1):22. doi: 10.1186/s12871-020-0941-1. PMID 31973700
- [Result] Akerman M, Pejcic N, Velickovic I. A Review of the Quadratus Lumborum Block and ERAS. Front Med (Lausanne). 2018 Feb 26;5:44. doi: 10.3389/fmed.2018.00044. eCollection 2018. PMID 29536008